CLINICAL TRIAL: NCT00168012
Title: An Open Study to Evaluate the Safety and Efficacy of IVIG-F10 in Patients With Primary Immunodeficiency Diseases (PID)
Brief Title: Efficacy and Safety of Intravenous Immunoglobulin IVIG-F10 in Patients With Primary Immunodeficiencies (PID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLB04_005CR
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Agammaglobulinemia; IgG Deficiency; Common Variable Immunodeficiency
Keywords: Immunoglobulin intravenous; Agammaglobulinemia; Hypogammaglobulinemia; Common variable immunodeficiency; Immunoglobulin G; Children
MeSH Terms: conditions — Agammaglobulinemia; IgG Deficiency; Common Variable Immunodeficiency | interventions — Immunoglobulins, Intravenous

INTERVENTIONS:
Drug: Immunoglobulins Intravenous (Human)

SUMMARY:
The purpose of this study is to demonstrate the effect of IVIG-F10 on the prevention of serious bacterial infections in patients with primary immunodeficiency.

As secondary endpoints the rate of overall infections, the tolerability and safety of IVIG-F10 are studied.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with primary immunodeficiency
* Regular IVIG therapy for at least 6 months prior to receiving IVIG-F10

Key Exclusion Criteria:

* Allergic reactions to immunoglobulins or other blood products
* Steroids (oral and parenteral, daily ≥0.15 mg of prednisone equivalent/kg/day
* History of cardiac insufficiency
* Epilepsia

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42
Dates: Start 2004-09; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Proportion of infusions temporally (during the infusion and within 48 hours after the end of infusion) associated with one or more adverse events, regardless of relationship.

SECONDARY OUTCOMES:
Rate of acute serious bacterial infections
Number of days out of work/school due to underlying PID
Number of infections
Rate, severity and relationship of all adverse events

REFERENCES:
- [Result] Berger M, Cunningham-Rundles C, Bonilla FA, Melamed I, Bichler J, Zenker O, Ballow M. Carimune NF Liquid is a safe and effective immunoglobulin replacement therapy in patients with primary immunodeficiency diseases. J Clin Immunol. 2007 Sep;27(5):503-9. doi: 10.1007/s10875-007-9096-9. Epub 2007 May 4. PMID 17479360